CLINICAL TRIAL: NCT05513677
Title: Characterisation of Biofilm Growth on Coated vs. Uncoated Urinary Catheter Surfaces in Normal Clinical Use
Acronym: PRO30CSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camstent Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRO30CSP
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: 1. Evaluated Patients: 5 patients (Convenience sample: non-blinded, non-randomised)
     Selection follows documented hospital protocols for routine catheterisation
  2. Measured Patients: 30 patients (Convenience sample: non-blinded and non-randomised)
     * 20 who receive the M4D coated catheter.
     * 10 who receive the standard uncoated catheters used in routine patient care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of Care
  Interventions: Device: Standard of Care
- M4D coated catheter (Experimental): Experimental
  Interventions: Device: M4D

INTERVENTIONS:
Device: M4D — Coated catheter
  Arms: M4D coated catheter
Device: Standard of Care — Standard of Care
  Arms: Standard of Care

SUMMARY:
1. Evaluated Patients: 5 patients (Convenience sample: non-blinded, non-randomised)

   Selection follows documented hospital protocols for routine catheterisation
2. Measured Patients: 30 patients (Convenience sample: non-blinded and non-randomised)

   * 20 who receive the M4D coated catheter.
   * 10 who receive the standard uncoated catheters used in routine patient care.

DETAILED DESCRIPTION:
1. Evaluated Patients: 5 patients (Convenience sample: non-blinded, non-randomised)

   Selection follows documented hospital protocols for routine catheterisation
2. Measured Patients: 30 patients (Convenience sample: non-blinded and non-randomised)

   * 20 who receive the M4D coated catheter.
   * 10 who receive the standard uncoated catheters used in routine patient care.

1) Evaluation (5 patients, coated catheter)

A convenience sample of patients will be selected to receive the Camstent coated catheter for their routine care. These enrolments are drawn from among those recommended for routine catheterisation, for up to 28 days and in accordance to existing hospital protocols. There is no change to the routine protocols for insertion, maintenance, withdrawal, or documentation of the patient's catheterisation. Following use, the catheter is discarded according to the hospital's procedures.

Staff questionnaires will be completed to capture general use information. These will document the opinions of the nurse inserting and withdrawing the catheter, and may include questions for the patient, to record their experience. There will be no collection of patient information, and no analysis of the discarded catheter.

2) Measurement (10 patients receiving uncoated catheters, 20 patients receiving coated catheters)

The data collection will include 10 patients who have received the standard hospital issued uncoated catheter and 20 patients who have received the Camstent coated catheter. There will be no randomisation and no blinding.

The first 10 patients needing routine urinary catheterisation to drain their bladder for up to 28 days whilst in hospital will receive the routine hospital issued catheter and will looked after by hospital and staff as standard practice.

The next 20 patients needing routine urinary catheterisation to drain their bladder whilst in hospital will receive a coated catheter. There will be no change to the intended use of the catheter for patients where it is deemed medically necessary to drain urine from the urinary bladder via the urethra using the catheter device for up to 28 days. There will be no change to any patient care or catheterisation procedures.

All 30 catheters will be sent to a laboratory for surface examination rather than immediately disposed of as medical waste. Harvested catheters will be bagged in an airtight plastic bag and tagged with a record identifier. A record identifier will be used to establish catheter traceability and duration, and will not compromise patient anonymity. The catheter will be kept refrigerated and transported to the analysis laboratory at Nottingham University within two days.

At the Nottingham Laboratory, the catheters will be subjected to qualitative and quantitative analysis to determine the percentage of biofilm coverage on the surface. This will initially be achieved using staining followed by microscopic visual examination of the catheter surface, and images taken of any surface encrustation.

For Fluorescence Microscopy, the procedure will be:

1. Cut the catheter into segments then wash three times in ~15 ml of PBS with gentle agitation.
2. Transfer the washed catheter segments into the wells of a sterile 24 well plate and stain with SYTO17 Red Fluorescent Nucleic Acid Stain.
3. Segments will be imaged using a laser scanning confocal microscope using a 10 X objective lens over a 1024 μm x 1024 μm area.
4. A z-section will be imaged (each section is 4μm apart with 36 images taken over 140μm) such that the entire curved surface is imaged. The coverage data will then be taken from a maximum intensity z-projection.
5. Data analysis will be carried out in ImageJ using the maximum intensity z-projection images.
6. Images will be converted to 8-bit greyscale images, a threshold applied to select the data correctly and the biofilm coverage measured.
7. The percentage of coverage for each sample will be computed as (Light) / (Light + Dark) * 100%.

Aggregate descriptive statistics will be calculated, and biofilm coverage will be plotted against the duration of catheterisation as a scattergram. The study is not powered to permit statistical analysis.

Prior laboratory experiments predict that the difference in biofilm coverage could exceed 80%. If larger differences are seen in harvested catheters, then a Total Cell Count assay, in which the biofilm is sonicated free of the surface and then assessed through serial dilution, may be substituted for Fluorescence Microscopy.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* • Patients under age 18.

  * Patients that have or recently (within 3 weeks) had a urinary catheter, or those with signs of current urinary tract infection.
  * Patients who they have had previous radiation therapy in lower pelvis.
  * Patients who are cognitively impaired, or are unwilling to give consent
  * Patients with a potentially immunocompromised condition
  * Patients that require further antibiotics after initial dose, or those that are administered antibiotics following an infection whilst the trial urinary catheter is in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the percentage of catheter surface colonised by biofilm, calculated as (light / (light + dark) x 100% in measurement of stained samples using fluorescence microscopy. | 30 days
  The primary outcome is the percentage of catheter surface colonised by biofilm, calculated as (light / (light + dark) x 100% in measurement of stained samples using fluorescence microscopy.

SECONDARY OUTCOMES:
Secondary outcomes will be logging of events, including catheter blockage or presumed CAUTI. | 30days
  Secondary outcomes will be logging of events, including catheter blockage or presumed CAUTI.

CONTACTS AND LOCATIONS:
Locations (1):
- The James Cook University Hospital,, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No